CLINICAL TRIAL: NCT02511314
Title: A Randomised, Controlled Trial of effectIveness of a Smart Sensor for Continence Care: the ARCTICC Study
Brief Title: A Trial of effectIveness of a Smart Sensor for Continence Care: the ARCTICC Study
Acronym: ARCTICC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: SCA Hygiene Products, AB (Unknown)
Responsible Party: Principal Investigator, Adrian Wagg, Research Chair in Healthy Aging, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: ARC-NH-1205
Record Dates: First submitted 2015-05-12; First posted 2015-07-30 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Urinary Incontinence
Keywords: Nursing homes; quasi-experimental; mixed methods; parallel study; urinary incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Tena Identifi is an integrated electronic monitoring system based upon a wearable continence pad which allows registration of resident's micturition patterns over a 72 hour period, allowing caregivers to construct an individualised continence care plan, including use of appropriate products.
  To create a voiding report, a resident wears the Identifi Sensor Wear with an attached Identifi Logger for three consecutive days (72 hours). The logger continuously logs the moisture status of the brief. The resulting data is sent to a server via 3 G signal where it is mapped onto a graph indicating voiding times and volumes.
  Interventions: Device: TENA Identifi
- Control Intervention (No Intervention): The control portion of the study is "usual care", defined as the routine practices and procedures, including continence assessment approach, prescribed in the nursing home unit or facility.

INTERVENTIONS:
Device: TENA Identifi — TENA Identifi
  Arms: Intervention

SUMMARY:
The purpose of this study is to compare the use of an electronic incontinence identification system with nursing home support (Tena Identifi) versus usual care on the quality, resource use and outcomes of continence care for older residents of nursing care homes.

DETAILED DESCRIPTION:
This is a prospective, quasi-experimental, controlled study with a mixed methods design with qualitative and quantitative components.

ELIGIBILITY:
Inclusion Criteria:

* Nursing homes: A facility which:

  * provides care for residents over the age of 65 years
  * has an existing policy for continence care
  * is registered with the appropriate Provincial authorities
  * engages in recording of the RAI- MDS v2.0
* Residents: Nursing home residents over the age of 65 requiring a continence assessment upon entry to the nursing home or requiring a reassessment because of either a change in clinical status or provincial requirement shall be eligible for entry

Exclusion Criteria:

* Residents

  * at the end of life,
  * with profound behavioural disturbances likely to render the use of the Tena Identifi system impractical
  * an identifiable, potentially reversible cause for their urinary incontinence (e.g.: acute urinary tract infection)
  * with double incontinence dominated by faecal incontinence
* Staff and Managers - Staff who did not take the training on the Identifi system or managers whose units that did not participate in the study will be ineligible for the focus group.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 89 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Between group change in the proportion of residents with a one category change in continence products usage | 8 weeks

SECONDARY OUTCOMES:
Between group change in time for construction of continence care plan following assessment | 8 weeks
Between group change in number of pads used | 8 weeks
Between group change in proportion of residents with pad leakage episodes | 8 weeks
Between group change in change in cost of continence products | 8 weeks
Between group change in change in healthcare aide / personal support worker time spent in continence care | 8 weeks
Between group change in Quality of life, measured by QoL AD | 8 weeks
Between group change in Activities of daily living as measured by Barthel index | 8 weeks
Between group change in number of wet checks at night | 8 weeks
Between group change in reduction in number of residents on "timed toileting schedules" | 8 weeks
Utility and acceptability of the Tena Identifi system by the end-user through a Focus Group | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Adrian S Wagg, MD, Principal Investigator — University of Alberta
Locations (1):
- Division of Geriatric Medicine, Clinical Sciences Building, University of Alberta Hosp, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Yu P, Hailey D, Fleming R, Traynor V. An exploration of the effects of introducing a telemonitoring system for continence assessment in a nursing home. J Clin Nurs. 2014 Nov;23(21-22):3069-76. doi: 10.1111/jocn.12538. Epub 2014 Jan 31. PMID 24479697
- [Background] Nikoletti S, Young J, King M. Evaluation of an electronic monitoring device for urinary incontinence in elderly patients in an acute care setting. J Wound Ostomy Continence Nurs. 2004 May-Jun;31(3):138-49. doi: 10.1097/00152192-200405000-00008. PMID 15867743
- [Background] Offermans MP, Du Moulin MF, Hamers JP, Dassen T, Halfens RJ. Prevalence of urinary incontinence and associated risk factors in nursing home residents: a systematic review. Neurourol Urodyn. 2009;28(4):288-94. doi: 10.1002/nau.20668. PMID 19191259
- [Background] Roe B, Flanagan L, Jack B, Shaw C, Williams K, Chung A, Barrett J. Systematic review of descriptive studies that investigated associated factors with the management of incontinence in older people in care homes. Int J Older People Nurs. 2013 Mar;8(1):29-49. doi: 10.1111/j.1748-3743.2011.00300.x. Epub 2011 Dec 19. PMID 22182302
- [Derived] Rajabali SN, Hunter KF, Asaana P, McCreary ML, Nazari S, Wagg AS. Effectiveness of a Smart Urinary Continence Care Assessment System for Nursing Home Residents: A Quasi-Experimental, Sequential Quantitative-Qualitative Methods Trial. J Wound Ostomy Continence Nurs. 2023 Jan-Feb 01;50(1):48-56. doi: 10.1097/WON.0000000000000937. PMID 36640164